CLINICAL TRIAL: NCT05655403
Title: Investigating the Effects of Step Training and the Mediating Effects of Prefrontal Cortex Functioning in Older Adults with Mild Dementia: a Randomized Wait-list Controlled Trial
Brief Title: Effects of Step Training in Older Adults with Mild Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: University Grants Committee, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr. Wayne Chan, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20221201007
Record Dates: First submitted 2022-12-02; First posted 2022-12-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Dementia
Keywords: Step training; Falls; Dementia; Randomized controlled trial; Prefrontal cortex
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Step training group (Experimental): The participants assigned to the ST condition will receive a 40-minute ST session twice a week for 12 weeks. The sessions will be delivered at community centers for older adults by an instructor with at least 5 years of experience in dementia care. Each session will consist of a 5-minute flexibility exercise warm-up, a 30-minute stepping exercise, and a 5-minute cool-down. A non-slip plastic mat marked with two standing panels and a number of removable stepping panels that can be secured to the plastic mat using hook-and-loop fasteners will be used as the exercise device. While standing on the standing panels, the participants will receive verbal instructions to (1) use one of their feet to step on a specific stepping panel and (2) return the stepping foot to the standing panel multiple times throughout every session.
  Interventions: Behavioral: Step training program
- Wait-list control group (Active Comparator): The participants assigned to the WC condition will then receive usual care for 12 weeks. After completing the 12-week assessment, they will complete the ST program.
  Interventions: Behavioral: Step training program

INTERVENTIONS:
Behavioral: Step training program — The program will consist of 3 phases: (1) getting familiar, (2) increasing complexity, and (3) consolidating skills. In Phase 1, the participants will be asked to use one foot to step on single-colored stepping panels located in a specific region of the plastic mat (e.g., upper quadrant). In Phase 2, the exercise will progress by introducing the following 4 cognitively challenging stepping tasks. After finishing the 4 stepping tasks in Phase 2, the exercises will progress to Phase 3, which will consolidate the participants' stepping and cognitive skills. The following 4 additional stepping tasks will be introduced. The instructor will tailor the exercises for each participant, based on their training performance.

SUMMARY:
Step training has been shown to be effective at reducing the incidence of falls and improving related risk factors, including choice stepping, in healthy older adults. However, the effects of step training have not been investigated in OWMD. The primary objective of the proposed project will be to assess the effects of a step-training program involving concurrent stepping and visuospatial tasks on choice stepping, prefrontal cortex functioning during choice stepping, and fall-related outcomes (i.e., step length, lower-limb muscle strength, balance, mobility, dual-task ability, and fear of falling) in OWMD.

The prefrontal cortex is responsible for the executive functions such as attention and inhibitory function, which are integral to choice stepping reaction time tasks. However, the effects of step training on prefrontal cortex functioning during choice stepping in OWMD remain unclear. The neural mechanisms underlying the potential effects of step training on choice stepping have never been investigated in this population. Therefore, the secondary objective of the proposed project will be to evaluate the mediating effects of changes in the prefrontal cortex functioning during choice stepping on the potential benefits of a step-training program for choice stepping in OWMD.

The proposed project will provide robust evidence to support the use of step training to improve choice stepping and reduce the risk of falls in OWMD. Disentangling the neural mechanisms underlying the effects of step training will be crucial to the development of the most effective interventions to target these mechanisms.

DETAILED DESCRIPTION:
Falls are common in older adults with mild dementia (OWMD), and they are the leading cause of functional dependence, morbidity, and mortality in this population. The ability to take rapid, accurate, and effective steps in varied environmental conditions, such as walking on a wet floor or rough terrain, is crucial to ensuring safety and avoiding falls. OWMD often have difficulties in choice stepping (i.e., stepping on a specific target, while avoiding irrelevant distractions), which requires high levels of sensorimotor and cognitive function. As impaired choice stepping has been shown to predict falls in the general older population, improving choice stepping is expected to reduce the risk of falls in OWMD.

Step training has been shown to be effective at reducing the incidence of falls and improving related risk factors, including choice stepping, in healthy older adults. However, the effects of step training have not been investigated in OWMD. The primary objective of the proposed project will be to assess the effects of a step-training program involving concurrent stepping and visuospatial tasks on choice stepping, prefrontal cortex functioning during choice stepping, and fall-related outcomes (i.e., step length, lower-limb muscle strength, balance, mobility, dual-task ability, and fear of falling) in OWMD.

The prefrontal cortex is responsible for the executive functions such as attention and inhibitory function, which are integral to choice stepping reaction time tasks. However, the effects of step training on prefrontal cortex functioning during choice stepping in OWMD remain unclear. The neural mechanisms underlying the potential effects of step training on choice stepping have never been investigated in this population. Therefore, the secondary objective of the proposed project will be to evaluate the mediating effects of changes in the prefrontal cortex functioning during choice stepping on the potential benefits of a step-training program for choice stepping in OWMD.

The proposed project will provide robust evidence to support the use of step training to improve choice stepping and reduce the risk of falls in OWMD. Disentangling the neural mechanisms underlying the effects of step training will be crucial to the development of the most effective interventions to target these mechanisms. Furthermore, the scientific evidence derived from the proposed project will motivate patients, caregivers, and clinicians to participate in such programs, and subsequently, relieve the fall-related burdens on multiple stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* at least 65 years old;
* have a physician's diagnosis of dementia according to the Diagnostic and Statistical Manual of Mental Disorders 5th edition;
* have mild dementia, indicated by a score of 10 or higher on the Montreal Cognitive Assessment Hong Kong version (HK-MoCA);
* able to walk 10 meters independently without a walking aid;
* receiving care by an unpaid "main caregiver" with at least 3.5 hours of face-to-face contact per week.

Exclusion Criteria:

* unable to perform step training due to unstable or severe musculoskeletal, cardiorespiratory, or neurological conditions;
* have severe hearing and/or visual impairments that limit their ability to communicate;
* have been hospitalized within the past 30 days.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Choice stepping reaction time test (CSRTT) | Post-intervention (week 12)
  Participants will be asked to stand on a non-slip plastic mat marked with two standing panels and four stepping panels. The RA will provide verbal instructions to (1) use one foot to step on a stepping panel to the front or the side and (2) return the stepping foot to the standing panel. The participants will complete 20 stepping trials as quickly as possible based on a fixed pre-determined sequence. The first 8 trials will be regarded as practice trials. The total time to complete the last 12 trials will be measured in seconds using a stopwatch.

SECONDARY OUTCOMES:
Prefrontal cortex (PFC) functioning during choice stepping | Post-intervention (week 12)
  fNIRS will be used to measure PFC activity during stepping tasks. Participants will be asked to stand on the same plastic mat used in the CSRTT. They will be asked to finish 2 rounds of stepping tasks, with 8 stepping blocks in each round and 8 stepping trials per block (i.e., active periods). The stepping performance of the participants will be videotaped using a handheld camera, and the number of correct and incorrect steps taken according to the verbal cues provided will be counted.
  Each stepping round will consist of 4 simple and 4 choice stepping blocks. In the simple stepping block, the participants will be verbally instructed to use the same foot to repeatedly step on the same panel. In the choice stepping block, they will be asked to use either the left or right foot to step on different panels in each trial.
Maximum step length test (MSLT) | Post-intervention (week 12)
  Participants will be asked to use their left or right foot to step 1) forward, (2) sideways, and (3) backward as far as they can without losing their balance. The mean distance covered in 5 stepping trials for each foot and direction will be recorded separately.
30-second sit-to-stand test (30STS) | Post-intervention (week 12)
  Participants will be asked to repeatedly rise from a chair and sit down. The number of repetitions completed in 30 seconds will be recorded.
Berg Balance Scale (BBS) | Post-intervention (week 12)
  The BBS consists of 14 items measuring the balance performance during daily functional activities, such as chair transfer, standing with eyes closed, turning 360 degrees, tandem standing, and single-leg standing. The total score ranges from 0 to 56, with a higher score indicating better balance.
Iconographical Fall Efficacy Scale - Chinese version (Icon-FES) | Post-intervention (week 12)
  The Icon-FES uses a combination of illustrations to assess concerns about falling during 10 daily activities, such as changing clothes, taking a shower, and changing a light bulb. The total score ranges from 0 to 40, with a higher score indicating a greater fear of falling.
Timed Up and Go Single Task (TUG-S) and Timed Up and Go Dual Task (TUG-D) | Post-intervention (week 12)
  In the TUG-S, the participants will be instructed to rise from an armchair, walk 3 meters, turn 180 degrees, walk back to the chair, and sit down at their own pace, and the time taken to complete the task will be recorded. For the TUG-D, the participants will be asked to perform the TUG-S while simultaneously naming as many animals as possible. The time used to complete the TUG-D and the dual-task cost (i.e., the time difference between the TUG-D and TUG-S) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne LS Chan, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No